CLINICAL TRIAL: NCT00461643
Title: Comparison of Three Different Strategies for Treating Infertility in Anovulatory Women With Polycystic Ovary Syndrome: a Multicentre Randomized Controlled Clinical Trial
Brief Title: Strategies for Ovulation Induction in Anovulatory Infertile Patients With PCOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01/2007
Record Dates: First submitted 2007-04-13; First posted 2007-04-18 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Anovulatory Infertility Related to Polycystic Ovary Syndrome
Keywords: Anovulation; Clomiphene citrate; Infertility; Metformin; PCOS; RCT; Treatment
MeSH Terms: conditions — Anovulation; Infertility | interventions — Clomiphene; Metformin; Gonadotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Strategy A (Active Comparator): clomiphene followed by clomiphene plus metformin followed by gonadotropins
  Interventions: Drug: Clomiphene citrate, metformin, metformin plus clomiphene citrate, gonadotropins
- Strategy B (Active Comparator): metformin followed by metformin plus clomiphene followed by gonadotropins
  Interventions: Drug: Clomiphene citrate, metformin, metformin plus clomiphene citrate, gonadotropins
- Strategy C (Active Comparator): metformin plus clomiphene followed by gonadotropins
  Interventions: Drug: Clomiphene citrate, metformin, metformin plus clomiphene citrate, gonadotropins

INTERVENTIONS:
Drug: Clomiphene citrate, metformin, metformin plus clomiphene citrate, gonadotropins

SUMMARY:
Anovulatory infertility is a common feature of the polycystic ovary syndrome (PCOS). Even if several first-step treatments have been proposed for anovulatory infertile PCOS patients, very few data are available in literature regarding the best integrated strategy. In fact, a single compound could be effective as first-step approach but not or less useful when integrated in a more complex strategy.

The goal of the current protocol will be to compare three different strategies for treating anovulatory infertility in PCOS patients having as primary end-point the multiple pregnancy rate.

DETAILED DESCRIPTION:
All patients eligible will undergo baseline assessment consisting of antropometric, hormonal, and ultrasonographic assessments. Successively, patients enrolled will be allocated in three different strategies (strategy A, B, and C).

A total of 184 infertile PCOS patients per arm will be enrolled and treated with three different integrated strategies: clomiphene followed by clomiphene plus metformin followed by gonadotropins (strategy A); metformin followed by metformin plus clomiphene followed by gonadotropins(strategy B); and metformin plus clomiphene followed by gonadotropins(strategy C).

In all patients, the same regimen will be used to administered clomiphene, metformin, and gonadotropins.Both clomiphene and metformin will be administered at incremental doses in each case.Gonadotropins will be administrated to obtain a controlled ovarian stimulation using highly purified urinary FSH in a low-dose step-up protocol.

During the study, the clinical and reproductive outcomes, and adverse experiences will be evaluated in each woman.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (using ESHRE/ARSM 2004 criteria)

Exclusion Criteria:

* Age <18 or >35 years
* Severe obesity (BMI >35)
* Neoplastic, metabolic, hepatic, and cardiovascular disorders or other concurrent medical illnesses
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia
* Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, antidiabetic and anti-obesity drugs or other hormonal drugs
* Previous use of ovulation induction agents
* Intention to start a diet or a specific program of physical activity
* No uterine bleeding after progesterone challenge test
* Organic pelvic diseases
* Previous pelvic surgery
* Suspected peritoneal factor infertility
* Tubal or male factor infertility or sub-fertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 552 (Estimated)
Dates: Start 2007-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Multiple pregnancy rate | 9 months

SECONDARY OUTCOMES:
Ovulation rate | 15 months
Pregnancy rate | 15 months
Abortion rate | 15 months
Live-birth rate | 24 months
Adverse-events | 15

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (2):
- Italy (2):
  - "Pugliese" Hospital, Catanzaro
  - Pugliese-Ciaccio Hospital, Catanzaro

REFERENCES:
- [Background] Palomba S, Orio F Jr, Falbo A, Manguso F, Russo T, Cascella T, Tolino A, Carmina E, Colao A, Zullo F. Prospective parallel randomized, double-blind, double-dummy controlled clinical trial comparing clomiphene citrate and metformin as the first-line treatment for ovulation induction in nonobese anovulatory women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Jul;90(7):4068-74. doi: 10.1210/jc.2005-0110. Epub 2005 Apr 19. PMID 15840746
- [Background] Moll E, Bossuyt PM, Korevaar JC, Lambalk CB, van der Veen F. Effect of clomifene citrate plus metformin and clomifene citrate plus placebo on induction of ovulation in women with newly diagnosed polycystic ovary syndrome: randomised double blind clinical trial. BMJ. 2006 Jun 24;332(7556):1485. doi: 10.1136/bmj.38867.631551.55. Epub 2006 Jun 12. PMID 16769748
- [Background] Legro RS, Barnhart HX, Schlaff WD, Carr BR, Diamond MP, Carson SA, Steinkampf MP, Coutifaris C, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Giudice LC, Leppert PC, Myers ER; Cooperative Multicenter Reproductive Medicine Network. Clomiphene, metformin, or both for infertility in the polycystic ovary syndrome. N Engl J Med. 2007 Feb 8;356(6):551-66. doi: 10.1056/NEJMoa063971. PMID 17287476